CLINICAL TRIAL: NCT02808559
Title: PASIMAT: Automatic Measure of PASI by Skin Imaging
Brief Title: PASIMAT: Automatic Measure of PASI
Acronym: PASIMAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: Pfizer (Industry); Fotofinder (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-AOI-01
Record Dates: First submitted 2016-06-15; First posted 2016-06-21 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bodystudio ATBM (Experimental): The PASI of the patients will be evaluated by two dermatologists then by the bodystudio ATBMs.
  Interventions: Device: Bodystudio ATBM (Automatic Total Body Mapping)

INTERVENTIONS:
Device: Bodystudio ATBM (Automatic Total Body Mapping) — The mapping of the entire body is automatically done using a high-resolution apparatus (20 photographs of the patient in 8 positions (face, back, lateral left and right, specific extremities) The photographs will be done with a standardized procedure established by FotoFinder. Every lesion is completely evaluated and the PASI score can be calculated.

SUMMARY:
To quantify the severity of psoriasis in a consistent and clinically meaningful way is important in order to decide the therapeutic orientation to take for the patient. PASI (Psoriasis Area and Severity Index) scoring is recognised as gold standard for psoriasis assessment. The bodystudio ATBM (Automatic Total Body Mapping) is a high-tech system performing standardized photos from head to feet and from all angles, which allows to map the entire skin covering all the human body in a few minutes.The primary objective of this study would be to evaluate the ability of the bodystudio ATBM to calculate the PASI score of patients with psoriasis human body in a few minutes

DETAILED DESCRIPTION:
Psoriasis is a chronic inflammatory skin condition resulting in a significant impact on patients' quality of life. To quantify the severity of psoriasis in a consistent and clinically meaningful way is important in order to decide the therapeutic orientation to take for the patient. PASI (Psoriasis Area and Severity Index) scoring is recognised as gold standard for psoriasis assessment. However the measure of the PASI score is very complex. Given this complexity, the PASI is influenced by inter and intra-rater variation. In addition the PASI assessment process is time consuming. The bodystudio ATBM (Automatic Total Body Mapping) is a high-tech system performing standardized photos from head to feet and from all angles, which allows to map the entire skin covering all the human body in a few minutes. The mapping of the entire body is automatically done by the use of a digital camera performing 20 pictures of the patient with 8 successive positions. The system is coupled to a software of automatic analysis of these pictures for the measure of the PASI score. The primary objective of this study would be to evaluate the ability of the bodystudio ATBM to calculate the PASI score of patients with psoriasis

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old
* Subject is affiliated to a National Health System at screening visit
* Understand and sign an Informed Consent Form (ICF) at screening, prior to any investigational procedures being performed.
* Patient with moderate to severe Plaque psoriasis.
* The patient is willing and able to be evaluated by the Bodystudio ATBM: 3 minutes for a young patient and until 7 minutes for an oldest.
* The patient is able to staying up during all the total body mapping procedure

Exclusion Criteria:

* The subject is vulnerable (such as deprived from freedom) as defined in Section 1.61 of International Conference on Harmonisation (ICH) Guideline for Good Clinical Practice (GCP).
* Pregnant woman or who are breast-feeding
* Patient with tattoos that could influence the PASI assessment.
* Patient with skin type (phototype) V or IV according to Fitzpatrick classification
* Male patients with exceeding facial or skin hair that could influence the automatic PASI assessment.
* Patients with exceeding varicose veins.
* Patients with sun burn

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index | one day

IPD SHARING:
Plan to Share IPD: Undecided